CLINICAL TRIAL: NCT02386267
Title: Therapeutic Use of the Amino Acid Leucine in the Treatment of Transfusion-Dependent Diamond Blackfan Anemia Patients
Brief Title: L-leucine in Diamond Blackfan Anemia Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Scientific Clinical Centre of Pediatric Hematology, Oncology and Immunology named after Dmitry Rogache (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ru0001
Record Dates: First submitted 2015-02-18; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Diamond Blackfan Anemia
MeSH Terms: conditions — Anemia, Diamond-Blackfan | interventions — Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-leucine pills (Experimental): L-leucine , dose- 700mg/m2 , per os, three time a day, course duration 6 months
  Interventions: Drug: L-leucine

INTERVENTIONS:
Drug: L-leucine — L-leucine pills per os for 6 months

SUMMARY:
Diamond-Blackfan anemia (DBA) is a rare congenital syndrome associated with physical anomalies, short stature, red cell aplasia, and an increased risk of malignancy.

Mutations affecting genes encoding ribosomal proteins cause DBA. Genetic studies have identified heterozygous mutations in at least one of eight ribosomal protein genes in up to 50% of cases.

25% of patients carry a mutation in the ribosomal protein (RP)S19 gene, whereas mutations in RPS24, RPS17, RPL35A, RPL11, and RPL5 are rare.

p53 activation has been identified as a key component in the pathophysiology of DBA after cellular and molecular studies. Other potential mechanisms that warrant further investigation include impaired translation as the result of ribosomal insufficiency, which may be ameliorated by Leucine supplementation.

Despite significant improvements in understanding of the pathophysiology of Diamond Blackfan anemia (DBA), there have been few advances in therapy. The cornerstones of treatment remain corticosteroids,chronic red blood cell transfusions, and hematopoietic stem cell transplantation, each of which is fraught with complications. Other treatments have been shown to be effective in only a few patients or in individual case reports : IL-3, cyclosporine (alone or in combination with steroids), metaclopramide. Gene therapy is still a part of research programs.

There are some indications that the Amino Acid (AA) L-leucine, a translation enhancer, may have some efficacy in DBA and 5q-syndrome, which has the same altered ribosome functions as the DBA. L-leucine is an essential AA that is unique among the branched-chain AA acting as a nutrient regulator of protein synthesis in skeletal muscle and adipose tissue.

Several preclinical studies with DBA lymphocytes exposed to various L-leucine doses, have demonstrated that protein synthesis can be increased by using high doses L-leucine.

Recent clinical data on L-leucine therapeutic use have demonstrated increase the hemoglobin level and transfusion independence in patients with DBA and 5q-syndrom.

These data support the rationale for clinical trial on L-leucine use as a therapeutic agent for DBA patients.

DETAILED DESCRIPTION:
Experimental: one arm L-leucine , dose- 700mg/m2 , per os, 3 time a day, 6 months

ELIGIBILITY:
Inclusion Criteria:

* signed Informed Consent Form
* diagnosed Diamond Blackfan Anemia
* transfusion dependenсe
* adequate renal function
* adequate liver function
* negative B-HCG and adequate contraception

Exclusion Criteria:

* known hypersensitivity to branched chain amino acids
* diagnosed AA metabolism disorder
* prior HSCT
* pregnancy or planning to become pregnant

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | every 4 weeks for 12 months
  Response to the treatment can be one of the following:
  1. Complete response (CR): Hb > 9 gm/dL and transfusion-independence as defined in DBA
  2. Partial response (PR): Hb < 9 gm/dL, increased reticulocyte count > 1% and any increase in transfusion interval from baseline.
  3. No response (NR): no change in transfusion requirements and no significant change in Hb or reticulocytes
  4. Progression: worsening of disease as defined by the need for more frequent transfusions

SECONDARY OUTCOMES:
Side effects of L-leucine in transfusion-dependent DBA patients for one year | every 4 weeks for 12 moths

CONTACTS AND LOCATIONS:
Overall Officials: Natalia - SMETANINA, MD, PhD, Principal Investigator — FSCCPHOI, Outpatient Department
Locations (1):
- Federal Scientific Clinical Centre of Pediatric Hematology Oncology Immunology n.a. Dmitry Rogachev, Moscow, Russia